CLINICAL TRIAL: NCT00860236
Title: Chronic Fatigue Syndrome and Abdominal Symptoms After Giardia Infection: Clinical Evaluation, Biomarkers, Risk Factors and the Effect of Intervention
Brief Title: Giardia Induced Fatigue and Functional Gastrointestinal Diseases
Acronym: GIFF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Nina Langeland, Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIFF
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Chronic Fatigue Syndrome
Keywords: CFS; Giardia; Fatigue; Cognitive behavioural therapy; CBT; Chronic fatigue syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Giardiasis; Fatigue | interventions — Counseling; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psycoeducation/counseling (Active Comparator)
  Interventions: Other: Psycoeducation/counseling
- Cognitive behavioural therapy (Active Comparator)
  Interventions: Behavioral: Cognitive behavioural therapy

INTERVENTIONS:
Other: Psycoeducation/counseling — 2 days of education on mechanisms of illness and coping strategies
  Arms: Psycoeducation/counseling
Behavioral: Cognitive behavioural therapy — 4 days intensive training in understanding and behavioural changes
  Other Names: CBT
  Arms: Cognitive behavioural therapy

SUMMARY:
A giardiasis outbreak in Bergen has given us the opportunity to approach two basic research questions of national and global importance:

* Studying the pathoimmunology of giardiasis in a natural setting, and following the genetic and immunological responses leading to recovery or persistent disease and sequelae.
* Studying the two disease entities FGID and CFS when induced by acute giardiasi and their risk factors.
* Interventional cognitive behavioural therapy is the only intervention documented to have significant effect on CFS outcome, and conventional cognitive behavioural therapy will be compared to a psycho-educational programme in the format of a randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Problems with fatigue of any severity after Giardia infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Improvement minimum 6 points in Chalder Fatigue scale score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bjarte Stubhaug, PhD, Study Director — Frihamnsenteret; Nina Langeland, PhD, Principal Investigator — University of Bergen
Locations (1):
- Frihamnsenteret, Skånevik, Norway